CLINICAL TRIAL: NCT03715699
Title: Leflunomide Treatment for IgG4-RD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Treatment for IgG4-RD
Record Dates: First submitted 2018-09-25; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Autoimmune Disease
MeSH Terms: conditions — Autoimmune Diseases | interventions — Prednisone; Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients treated with single glucocorticoid
  Interventions: Drug: Prednisone; Drug: Prednisone and Leflunomide
- Group 2 (Experimental): Patients treated with Leflunomide and glucocorticoid
  Interventions: Drug: Prednisone; Drug: Prednisone and Leflunomide

INTERVENTIONS:
Drug: Prednisone — Prednisone: started with prednisone alone 0. 6-0. 8mg/kg.d for 1 month, decreased 5mg per 2 weeks, and maintained at 7.5mg to 10mg/d to 12 months.
Drug: Prednisone and Leflunomide — Prednisone: started with prednisone 0. 6-0. 8mg/kg.d for 1 month, decreased 5mg per 2 weeks, maintained at 7.5mg to 10mg/d to 12 months.
  Leflunomide: 20mg qd for 6 months and 10mg qd for 6 months.

SUMMARY:
This study is an open-label randomized controlled trial aiming to investigate whether the efficacy and side effect of Leflunpomide plus glucocorticoid.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged 18 to 70 years old with informed consent
* All patients must meet the following diagnostic criteria of IgG4RD (2011):

  1. swelling, sclerosing and inflammatory involvement of one or more organ, including sclerosing pancreatitis, sialadenitis (Mikulicz disease), sclerosing cholangitis, inflammatory pseudotumors, retroperitoneal or mediastinal fibrosis, interstitial nephritis, hypophysitis, sclerosing dacryoadenitis, inflammatory aortic aneurysm, lymphadenopathy, or other inflammatory conditions;
  2. elevated serum IgG4 (>1.35 g/L);
  3. histopathologic features of fibrosis and/or lymphocytic and polyclonal plasma cell infiltration (and IgG4+ plasma cells on immunohistology when performed). Patients fulfill 1)+2)+3) are diagnosed as definite IgD4RD, 1)+2): possible IgG4RD; 1)+3): probable IgG4RD;
  4. exclusion of other diseases.

Exclusion Criteria:

* Patients will not be included if meets any of the following criteria:

  1. Patients who were diagnosed as other autoimmune diseases;
  2. Patients who were diagnosed as malignant diseases;
  3. Pregnant and lactating women；
  4. Active infection: HIV, HCV, HBV, TB；
  5. Serious organ function failure, expected life time less than 6 months.
  6. Presenting with Mikulicz disease without other manifestations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Response of Leflunomide treatment for IgG4-RD | 1 year
  Complete response rate; Partial response rate; No response

SECONDARY OUTCOMES:
Relapse of Leflunomide treatment for IgG4-RD | 1 year
  Clinical relapse; Serological relapse

CONTACTS AND LOCATIONS:
Locations (1):
- Yunyun Fei, Beijing, Beijing Municipality, China